CLINICAL TRIAL: NCT04235842
Title: Effects of Physical Exercise in Postoperative Bariatric Surgery Patients
Brief Title: Physical Exercise in Postoperative Bariatric Surgery Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, bariatric surgeries has been suspended and the center where the study was being developed still did not resume the bariatric surgeries. It is supposed to resume this year.
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Antonio Roberto Zamunér, Adjunct Professor - Principal Investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 284/2019
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Physical Exercise; Bariatric Surgery; Morbid Obesity
MeSH Terms: conditions — Motor Activity; Obesity, Morbid | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, single blinded.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the study intervention the participants were submitted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (No Intervention): The CG will receive the standard indications routinely provided by the hospital which consists in information about practice of regular physical activity according to World Health Organization. A leaflet with illustrations and indications will be provided and will be explained by the principal investigator.
- Moderate-intensity continuous exercise training group (GMICT) (Experimental): The GMICT will be submitted to a physical exercise program in which the aerobic component will be a moderate-intensity continuous exercise training, performed at 60% of the heart rate reserve, two days a week, for 30 minutes.
  Interventions: Other: Physical Exercise
- High-intensity interval training exercise group (GHIIT) (Experimental): The GHIIT will be will be submitted to a physical exercise program in which the aerobic component will be a high-intensity interval exercise training, performed in a protocol consisted of four one-min sprint at 90% of the heart rate reserve, alternated with one-min rest (at week 1) and progressing until reach 10 bouts of one-min sprint alternated with one-min rest.
  Interventions: Other: High-intensity interval training performed at cycle ergometer.

INTERVENTIONS:
Other: Physical Exercise — Moderate-intensity continuous exercise training performed at cycle ergometer.
  Arms: Moderate-intensity continuous exercise training group (GMICT)
Other: High-intensity interval training performed at cycle ergometer. — High-intensity interval training performed at cycle ergometer.
  Arms: High-intensity interval training exercise group (GHIIT)

SUMMARY:
This study aims to determine the effect of two types of exercise training on body composition, cardiopulmonary function and quality of life in people after undergoing bariatric surgery.

DETAILED DESCRIPTION:
Three groups will be studied:

1. Control group (CG)
2. Group of moderate intensity continuous aerobic exercise (GMICT)
3. High intensity interval aerobic exercise group (GHIIT)

The CG will follow the usual protocol adopted by the hospital San Juan de Dios, Curicó, Chile. The protocol consists in delivering information about relevance of engage in regular physical exercise practice according to the World Health Organization (150 minutes of activity per week moderate physical or at least 75 minutes of intense physical activity), but do not include the patients in a supervised physical exercise program.

The GMICT will undergo a physical exercise program in which the aerobic component will be a moderate-intensity continuous exercise training (60% of the heart rate reserve).

The GHIIT will undergo the same exercise program of the GMICT, but the aerobic component will be a high-intensity interval exercise training (10 sets of 1 min at 90% of heart rate reserve, with 1 min of rest between sets).

All groups will receive a nutritional diet plan prescribed by a specialist bariatric nutritionist blinded to the participants group assignment.

At the end of the study, the CG will be invited to enjoy the exercise program showing to be more effective.

Outcomes will be assessed at four time points: 1) one week before surgery; 2) 21 days after surgery (baseline before start exercise program); 3) 8 weeks after the beginning of the exercise program; and 4) one week after the end of intervention.

Main outcomes are: 1) body composition; 2) heart rate variability; 3) six-minute walk test and 4) quality of life. Secondary outcomes will be: 1) maximal respiratory pressures; 2) flowmeter; 3) dynamometry of upper limb; and 4) squat test in 30 seconds.

All procedures will be performed in the Hospital of Curicó, Chile, at the Department of Physical Medicine and Rehabilitation Service.

ELIGIBILITY:
Inclusion Criteria:

* Persons between 18 and 65 years old, both sexes, who have undergone bariatric surgery, with medical authorization to perform physical exercise, that the wound healing process operative is in the final phase, which have been administered with subsequent anti thrombus treatment to surgery, who have no plans to change their place of residence within the current year.

Exclusion Criteria:

* Persons who have had immediate complications after bariatric surgery (dehiscence anastomosis and operative wound dehiscence), presented any comorbidity decompensation after surgery, who are in the process of dialysis or who suffer from neuromotor disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body fat (%) | 16 weeks
  To determine the effects of HIIT and MCIT on body composition by measuring percent of body fat using a tetrapolar bioelectrical impedance.
Muscle mass (Kg) | 16 weeks
  To determine the effects of HIIT and MCIT on body composition by measuring muscle mass using a tetrapolar bioelectrical impedance.
Bone mass (Kg) | 16 weeks
  To determine the effects of HIIT and MCIT on body composition by measuring bone mass using a tetrapolar bioelectrical impedance.
Heart rate variability | 16 weeks
  To determine the effects of HIIT and MCIT on cardiac autonomic control in supine and orthostatic positions.
Six minutes walk test (mts traveled) | 16 weeks
  To determine the effects of HIIT and MCIT on functional capacity using the six-minute walk test.
Moorehead-Ardelt Quality of Life Questionnaire (MAQ II) | 16 weeks
  To determine the effects of HIIT and MCIT on quality of life by the Moorehead-Ardelt Quality of Life Questionnaire. The score of each answer ranges from -0.5 (most unfavorable situation) to +0.5 (most favorable situation). According to the score obtained: -3 to -2.1: "very poor"; -2 to -1.1: "poor"; -1 to 1: "fair"; 1.1 to 2: "good"; and 2.1 to 3: "very good" quality of life.
Bariatric Analysis and Reporting Outcomes System (BAROS Score) | 16 weeks
  To determine the effects of HIIT and MCIT on quality of life by the Bariatric Analysis and Reporting Outcomes System. Moorehead-Ardelt questionnaire incorporates the percentage of overweight lost or gained after surgery, resolution of comorbidities associated with morbid obesity, need for reoperation and complications. According to the score obtained, it is categorized as: ≤1: "failure"; > 1 to 3: "fair"; > 3 to 5: "good"; > 5 to 7: "very good"; and > 7 to 9: excellent.

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressures (cmH2O) | 16 weeks
  To determine the effects of HIIT and MCIT on the maximal inspiratory and expiratory pressures.
Flowmeter (L/min) | 16 weeks
  To determine the effects of HIIT and MCIT on the peak expiratory flow.
Hand grip strength test (Kg) | 16 weeks
  To determine the effects of HIIT and MCIT on the maximum prehensile force will be measured.
30-sec chair stand test (count) | 16 weeks
  To determine the effects of HIIT and MCIT on cardiopulmonary function the number of squats in 30 seconds will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Zamunér, PhD, Study Director — Universidad Católica del Maule
Locations (1):
- Hospital San Juan de Dios de Curicó, Curicó, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy, data will be stored and coded. At the end of the study, data may be available upon a reasonable request and ensuring the participants' data confidentiality will be preserved.

REFERENCES:
- [Background] Alcaraz Garcia AM, Ferrer Marquez M, Parron Carreno T. [Quality of life in obese patients and change after bariatric surgery medium and long term]. Nutr Hosp. 2015 May 1;31(5):2033-46. doi: 10.3305/nh.2015.31.5.8792. Spanish. PMID 25929372
- [Background] Amaya Garcia MJ, Vilchez Lopez FJ, Campos Martin C, Sanchez Vera P, Pereira Cunill JL. [Micronutrients in bariatric surgery]. Nutr Hosp. 2012 Mar-Apr;27(2):349-61. doi: 10.1590/S0212-16112012000200004. Spanish. PMID 22732956
- [Background] Carrasco F, Klaassen J, Papapietro K, Reyes E, Rodriguez L, Csendes A, Guzman S, Hernandez F, Pizarro T, Sepulveda A. [A proposal of guidelines for surgical management of obesity]. Rev Med Chil. 2005 Jun;133(6):699-706. doi: 10.4067/s0034-98872005000600013. Epub 2005 Jul 22. Spanish. PMID 16075135
- [Background] Brzozowska MM, Sainsbury A, Eisman JA, Baldock PA, Center JR. Bariatric surgery, bone loss, obesity and possible mechanisms. Obes Rev. 2013 Jan;14(1):52-67. doi: 10.1111/j.1467-789X.2012.01050.x. Epub 2012 Oct 25. PMID 23094966
- [Background] Carrasco F, Papapietro K, Csendes A, Salazar G, Echenique C, Lisboa C, Diaz E, Rojas J. Changes in resting energy expenditure and body composition after weight loss following Roux-en-Y gastric bypass. Obes Surg. 2007 May;17(5):608-16. doi: 10.1007/s11695-007-9117-z. PMID 17658019
- [Background] Cocks M, Shaw CS, Shepherd SO, Fisher JP, Ranasinghe A, Barker TA, Wagenmakers AJ. Sprint interval and moderate-intensity continuous training have equal benefits on aerobic capacity, insulin sensitivity, muscle capillarisation and endothelial eNOS/NAD(P)Hoxidase protein ratio in obese men. J Physiol. 2016 Apr 15;594(8):2307-21. doi: 10.1113/jphysiol.2014.285254. Epub 2015 Feb 24. PMID 25645978
- [Background] Coleman KJ, Caparosa SL, Nichols JF, Fujioka K, Koebnick C, McCloskey KN, Xiang AH, Ngor EW, Levy SS. Understanding the Capacity for Exercise in Post-Bariatric Patients. Obes Surg. 2017 Jan;27(1):51-58. doi: 10.1007/s11695-016-2240-y. PMID 27229736
- [Background] De Tursi Rispoli L, Vazquez Tarragon A, Vazquez Prado A, Saez Tormo G, Mahmoud Ismail A, Gumbau Puchol V. [Oxidative stress; a comparative study between normal and morbid obesity group population]. Nutr Hosp. 2013 May-Jun;28(3):671-5. doi: 10.3305/nh.2013.28.3.6355. Spanish. PMID 23848087
- [Background] Delgado Floody P, Cofre Lizama A, Alarcon Hormazabal M, Osorio Poblete A, Caamano Navarrete F, Jerez Mayorga D. [EVALUATION OF A COMPREHENSIVE PROGRAM OF FOUR MONTHS OF DURATION ON THE PREOPERATIVE CONDITIONS OF OBESE PATIENTS CANDIDATES FOR BARIATRIC SURGERY]. Nutr Hosp. 2015 Sep 1;32(3):1022-7. doi: 10.3305/nh.2015.32.3.9350. Spanish. PMID 26319815
- [Background] Delgado Floody P, Jerez Mayorga D, Caamano Navarrete F, Concha Diaz M, Ovalle Elgueta H, Osorio Poblete A. [EFFECTIVENESS OF COMPREHENSIVE TREATMENT ON THE PREOPERATIVE CONDITIONS OF OBESE WOMEN CANDIDATES FOR BARIATRIC SURGERY]. Nutr Hosp. 2015 Dec 1;32(6):2570-5. doi: 10.3305/nh.2015.32.6.9761. Spanish. PMID 26667705
- [Background] Delgado Floody P, Jerez Mayorga D, Caamano Navarrete F, Osorio Poblete A, Thuillier Lepeley N, Alarcon Hormazabal M. [TWELVE WEEKS OF PHYSICAL EXERCISE INTERVAL WITH SURCHARGE IMPROVES THE ANTHROPOMETRIC VARIABLES OF OBESE MORBID AND OBESE WITH COMORBIDITIES CANDIDATES TO BARIATRIC SURGERY]. Nutr Hosp. 2015 Nov 1;32(5):2007-11. doi: 10.3305/nh.2015.32.5.9610. Spanish. PMID 26545654
- [Background] Delgado Floody P, Caamano Navarrete F, Jerez Mayorga D, Campos Jara C, Ramirez Campillo R, Osorio Poblete A, Alarcon Hormazabal M, Thuillier Lepeley N, Saldivia Mansilla C. [Effects of a multidisciplinary program on morbid obese patients and patients with comorbility who are likely to be candidates for bariatric surgery]. Nutr Hosp. 2015 May 1;31(5):2011-6. doi: 10.3305/nh.2015.31.5.8569. Spanish. PMID 25929369
- [Background] Delgado Floody P, Caamano Navarrete F, Ovalle Elgueta H, Concha Diaz M, Jerez Mayorga D, Osorio Poblete A. Efectos de un programa de ejercicio fisico estructurado sobre los niveles de condicion fisica y el estado nutricional de obesos morbidos y obesos con comorbilidades. Nutr Hosp. 2016 Mar 25;33(2):107. doi: 10.20960/nh.107. Spanish. PMID 27238789
- [Background] Delgado Floody P, Caamano Navarrete F, Osorio Poblete A, Jerez Mayorga D. Variaciones en el estado nutricional, presion arterial y capacidad cardiorrespiratoria de obesos candidatos a cirugia bariatrica: beneficios del ejercicio fisico con apoyo multidisciplinar. Nutr Hosp. 2016 Feb 16;33(1):16. doi: 10.20960/nh.v33i1.16. Spanish. PMID 27019243
- [Background] Folope V, Chapelle C, Grigioni S, Coeffier M, Dechelotte P. Impact of eating disorders and psychological distress on the quality of life of obese people. Nutrition. 2012 Jul;28(7-8):e7-e13. doi: 10.1016/j.nut.2011.12.005. Epub 2012 Apr 7. PMID 22484005
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Guiraud T, Nigam A, Gremeaux V, Meyer P, Juneau M, Bosquet L. High-intensity interval training in cardiac rehabilitation. Sports Med. 2012 Jul 1;42(7):587-605. doi: 10.2165/11631910-000000000-00000. PMID 22694349
- [Background] Herring LY, Stevinson C, Carter P, Biddle SJH, Bowrey D, Sutton C, Davies MJ. The effects of supervised exercise training 12-24 months after bariatric surgery on physical function and body composition: a randomised controlled trial. Int J Obes (Lond). 2017 Jun;41(6):909-916. doi: 10.1038/ijo.2017.60. Epub 2017 Mar 6. PMID 28262676
- [Background] Hewitt S, Sovik TT, Aasheim ET, Kristinsson J, Jahnsen J, Birketvedt GS, Bohmer T, Eriksen EF, Mala T. Secondary hyperparathyroidism, vitamin D sufficiency, and serum calcium 5 years after gastric bypass and duodenal switch. Obes Surg. 2013 Mar;23(3):384-90. doi: 10.1007/s11695-012-0772-3. PMID 23015268
- [Background] Jung ME, Bourne JE, Beauchamp MR, Robinson E, Little JP. High-intensity interval training as an efficacious alternative to moderate-intensity continuous training for adults with prediabetes. J Diabetes Res. 2015;2015:191595. doi: 10.1155/2015/191595. Epub 2015 Mar 30. PMID 25918728
- [Background] Kessler HS, Sisson SB, Short KR. The potential for high-intensity interval training to reduce cardiometabolic disease risk. Sports Med. 2012 Jun 1;42(6):489-509. doi: 10.2165/11630910-000000000-00000. PMID 22587821
- [Background] Lund MT, Hansen M, Wimmelmann CL, Taudorf LR, Helge JW, Mortensen EL, Dela F. Increased post-operative cardiopulmonary fitness in gastric bypass patients is explained by weight loss. Scand J Med Sci Sports. 2016 Dec;26(12):1428-1434. doi: 10.1111/sms.12593. Epub 2015 Dec 4. PMID 26635069
- [Background] Matsuo T, Saotome K, Seino S, Shimojo N, Matsushita A, Iemitsu M, Ohshima H, Tanaka K, Mukai C. Effects of a low-volume aerobic-type interval exercise on VO2max and cardiac mass. Med Sci Sports Exerc. 2014 Jan;46(1):42-50. doi: 10.1249/MSS.0b013e3182a38da8. PMID 23846165
- [Background] Moorehead MK, Ardelt-Gattinger E, Lechner H, Oria HE. The validation of the Moorehead-Ardelt Quality of Life Questionnaire II. Obes Surg. 2003 Oct;13(5):684-92. doi: 10.1381/096089203322509237. PMID 14627461
- [Background] Papapietro K, Massardo T, Riffo A, Diaz E, Araya AV, Adjemian D, Montesinos G, Castro G. [Bone mineral density disminution post Roux-Y bypass surgery]. Nutr Hosp. 2013 May-Jun;28(3):631-6. doi: 10.3305/nh.2013.28.3.6400. Spanish. PMID 23848081
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Tschentscher M, Eichinger J, Egger A, Droese S, Schonfelder M, Niebauer J. High-intensity interval training is not superior to other forms of endurance training during cardiac rehabilitation. Eur J Prev Cardiol. 2016 Jan;23(1):14-20. doi: 10.1177/2047487314560100. Epub 2014 Nov 17. PMID 25404752
- [Background] Sim AY, Wallman KE, Fairchild TJ, Guelfi KJ. High-intensity intermittent exercise attenuates ad-libitum energy intake. Int J Obes (Lond). 2014 Mar;38(3):417-22. doi: 10.1038/ijo.2013.102. Epub 2013 Jun 4. PMID 23835594
- [Derived] Herrera-Santelices A, Tabach-Apraiz A, Andaur-Caceres K, Zamuner AR. Effect of physical exercise in bariatric surgery patients: protocol of a randomized controlled clinical trial. Trials. 2021 Feb 1;22(1):107. doi: 10.1186/s13063-021-05056-4. PMID 33522950
- See also: Selection of candidates for bariatric surgery — https://doi.org/10.1016/S0009-739X(04)72308-8
- See also: Epidemiology of obesity in Chile — https://doi.org/10.1016/S0716-8640(12)70287-0
- See also: Historias de vida: una metodología de investigación cualitativa. — https://revistas.upr.edu/index.php/griot/article/view/1775
- See also: Recomendaciones de la SECO para la práctica de la cirugía bariátrica y metabólica — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=2ahUKEwjo2_X7ivrmAhUcK7kGHcCGDGwQFjAAegQIBRAC&url=https%3A%2F%2Fwww.bmi-journal.com%2Findex.php%2Fbmi%2Farticle%2Fdownload%2F299%2Fpdf&usg=AOvVaw0fG0lZzYS_PxPl5PxiRc8R
- See also: ¿Cómo analizar datos cualitativos?. — http://www.ub.edu/ice/recerca/pdf/ficha7-cast.pdf
- See also: Evaluación mediante score BAROS de los resultados del bypass gástrico en el tratamiento de la obesidad mórbida — http://dx.doi.org/10.4067/S0718-40262006000500010
- See also: Alteraciones hepáticas en el paciente con obesidad mórbida sometido a cirugía bariátrica — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=4&ved=2ahUKEwjr9NPVi_rmAhVjFLkGHeKaASgQFjADegQIBhAB&url=https%3A%2F%2Fmedicinainterna.org.mx%2Farticle%2Falteraciones-hepaticas-en-el-paciente-con-obesidad-morbida-sometido-a-cirugia-bariatrica%2F&usg=AOvVaw37qDW5Feu0lMuLLudMrwCq
- See also: Tratamiento con cirugía bariátrica en el paciente obeso. — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=2ahUKEwi-i_78kPrmAhU_ILkGHXXkBN0QFjAAegQIBhAB&url=http%3A%2F%2Fve.scielo.org%2Fscielo.php%3Fscript%3Dsci_arttext%26pid%3DS1690-31102015000100007&usg=AOvVaw0HEowMfxGoTQKPxKKBDzh1
- See also: Encuesta Nacional De Salud 2016-2017, primeros resultados — https://www.minsal.cl/wp-content/uploads/2017/11/ENS-2016-17_PRIMEROS-RESULTADOS.pdf
- See also: Nota Descriptiva Obesidad y Sobrepeso — http://www.who.int/mediacentre/factsheets/fs311/es/
- See also: Exercise reduces lean mass loss in obese patients undergoing bariatric surgery — http://dx.doi.org/10.1016/j.rchic.2016.05.007
- See also: Evaluation of a structured program of physical exercise in morbidly obese patients awaiting bariatric surgery — http://dx.doi.org/10.3305/nh.2014.29.1.6937
- See also: Quality of life: A theoretical review — http://dx.doi.org/10.4067/S0718-48082012000100006
- See also: BODY COMPOSITION ASSESSMENT IN SPORTS MEDICINE. STATEMENT OF SPANISH GROUP OF KINANTHROPOMETRY OF SPANISH FEDERATION OF SPORTS MEDICINE — http://www.femede.es/documentos/ConsensoCine131.pdf